CLINICAL TRIAL: NCT00675064
Title: Single-blind, Placebo-controlled, Randomized Study Testing Single Ascending Doses of GSK369796 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ISO105774
Record Dates: First submitted 2008-04-22; First posted 2008-05-08 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Malaria
Keywords: pharmacokinetics,; safety; single ascending dose,; Healthy volunteers,
MeSH Terms: conditions — Malaria | interventions — N-tert-butylisoquine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anti-malarial experimental drug (Experimental): After randomization subjects will receive either 5, 25, 100, 250, 500, 1000, 2000 and 3000 mg of GSK3697969 orally . GSK3697969 will be available as 5, 25 and 250 mg capsules.
  Interventions: Drug: GSK369796
- Matching placebo (Active Comparator): After randomization subjects will receive matching placebo of GSK3697969.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK369796 — Anti-malarial
  Arms: Anti-malarial experimental drug
Drug: Placebo — Placebo matching GSK369796
  Arms: Matching placebo

SUMMARY:
This study will examine safety of single doses of GSK369796 in healthy subjects, along with some test to examine how quickly GSK369796 gets in your blood, and how long it takes your body to get rid of it.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between the ages of 18 to 40, inclusive.
* Female subjects must be of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or bilateral oophrectomy or postmenopausal defined as 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/ml.
* Body weight > 50 kg and body mass index (BMI) between 19 and 30 kg/m2 where:
* A screening electrocardiogram (12-lead ECG) with QTc <450 msec.
* Troponin I £0.04 ng/mL at screening with Beckman Access2® AccuTnI™ Troponin I Assay.
* The subject is able to understand and comply with protocol requirements, instructions and restrictions.
* Signed and dated written informed consent prior to admission to the study
* Healthy adult males and females between 18 and 60 years of age, inclusive. Whether a subject is "healthy" will be determined by a responsible physician, based on a medical evaluation including history, physical examination, laboratory tests, cardiac monitoring.
* To be eligible, female subjects must have a negative pregnancy test (i.e. serum bhCG test) and be of:

  1. non-childbearing potential (i.e. physiologically incapable of becoming pregnant). This includes pre-menopausal females with documented (medical report verification) hysterectomy or double oophrectomy or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy, or documented hysterectomy - tubal ligation is not sufficient.
  2. childbearing potential and agrees to commit to two of the protocol-approved methods of contraception, when used consistently and in accordance with both the product label and the instructions of a physician (and as listed in protocol).
* Male subjects must agree to abstain from or use a condom during sexual intercourse with pregnant or lactating females; or use a condom/spermicide, in addition to having their female partner use another form of contraception, such as an IUD, diaphragm with spermicide, oral contraceptive, inject able progesterone, or sub dermal implant if engaging in sexual intercourse with a female partner who could become pregnant. This criterion must be followed from the time of the first dose of study medication until completion of follow up procedures.
* Body weight ³ 50 kg (110 pounds) for men and ³ 45 kg (99 pounds) for women and body mass index (BMI) between 19 and 31.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and bilirubin within reference range at screening.
* Signed and dated written informed consent prior to admission to the study. The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening history and physical exam, screening 12-lead surface electrocardiogram (ECG), and screening 24-holter cardiac monitoring.
* Any evidence of cardiac disease or other clinically relevant abnormality identified on the screening echocardiography.
* Any clinically relevant abnormality on the clinical safety laboratory tests at screening.
* Positive for Human Immunodeficiency Virus (HIV) antibody, hepatitis B virus surface antigen, or hepatitis C virus antibody at screening.
* Significant cardiac history including but not limited to history of myocardial infarction, angina, heart failure, cardiomyopathy, arrhythmia, myocarditis, hypertrophy (atrial or ventricular), or cor pulmonale.
* Significant central nervous system (e.g., seizures), pulmonary, metabolic, renal, hepatic or gastrointestinal conditions or history of such conditions that, in the opinion of the investigator and/or GSK medical monitor, places the subject at an unacceptable risk as a participant in this trial or may interfere with the absorption, distribution, metabolism or excretion of drugs.
* History of sensitivity to any of the study medications or components thereof.
* History of sensitivity to 4-aminoquinolines (e.g., chloroquine, amodiaquine, or piperaquine).
* History of sensitivity to heparin or heparin-induced thrombocytopenia, if the clinical research unit will use heparin to maintain intravenous cannula patency.
* Use of prescription or non-prescription drugs, vitamins, herbal and dietary supplements within 14 days or 5 half-lives (whichever is longer) prior to study medication administration, or use of St. John's Wort within 28 days prior to the study medication administration Unless in the opinion of the investigator and sponsor the medication will not interfere with study procedures or compromise safety. By exception, the volunteer may take paracetamol (</ 2 grams/day) up to 48 hours prior to the study medication administration.
* Consumption of grapefruit, grapefruit juice, orange juice or Seville oranges, red wine within 7 days prior to administration of study medication.
* Participation in a clinical study of an investigational or non-investigational drug within 3 months or 5 half-lives (whichever is longer) preceding the study medication administration.
* Exposure to more than four new chemical entities within 12 months prior to dosing.
* History of drug abuse within 6 months of the study.
* A positive urine test for drugs of abuse or alcohol (or alcohol breath test) at screening or predose.
* History of smoking or use of nicotine containing products within 3 months of screening, or a positive urine cotinine indicative of smoking at screening.
* History of regular alcohol consumption exceeding 14 units/week or 2 units/day for women, or 21 units/week or 3 units/day for men, within 6 months of screening. One unit is equivalent to a half-pint of beer or 1 measure of spirits or 1 glass of wine.
* An unwillingness of male subjects to abstain from sexual intercourse with pregnant or lactating women, or an unwillingness of male subjects to use a condom/spermicide, in addition to having their female partner use another form of contraception such as an IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation, if engaging in sexual intercourse with a female partner who could become pregnant. This criterion must be followed from the time of study medication administration and until 84 days later.
* Donation of blood in excess of 500 mL within 90 days prior to dosing.
* An unwillingness to comply with lifestyle and/or dietary restrictions

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2008-05-02 (Actual); Primary Completion 2008-10-12 (Actual); Study Completion 2008-10-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | From Day 1 to follow-up visit

SECONDARY OUTCOMES:
Pharmacokinetics | Day 1 to Day 4

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: Results for study ISO105774 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/ISO105774?search=study&search_terms=ISO105774#rs